CLINICAL TRIAL: NCT01969058
Title: A Prospective Randomized Controlled Study to Evaluate the Effect of Isotretinoin on Immune Activation Among HIV-1 Infected Subjects With Incomplete CD4+ T Cell Recovery on Suppressive Antiretroviral Therapy (ART)
Brief Title: Effect of Isotretinoin on Immune Activation Among HIV-1 Infected Subjects With Incomplete CD4+ T Cell Recovery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5325; UM1AI068636 (NIH)
Record Dates: First submitted 2013-08-21; First posted 2013-10-25 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: HIV-1 Infection
Keywords: Isotretinoin; HIV-1; immunology markers; immune activation; viral suppression
MeSH Terms: interventions — Isotretinoin

STUDY DESIGN:
Intervention Model Description: Participants were randomized 2:1 to Isotretinoin arm and no study treatment arm. The primary endpoints were compared between the 2 study arms.
Masking Description: open label
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isotretinoin Arm (Active Comparator): Participants received Isotretinoin at approximately 0.5 mg/kg orally once daily for 4 weeks, then increased to approximately 1.0 mg/kg orally once daily for 12 weeks.
  Interventions: Drug: Isotretinoin
- No study treatment Arm (No Intervention): No Isotretinoin treatment

INTERVENTIONS:
Drug: Isotretinoin — Isotretinoin is a drug that is approved for use in the treatment of severe acne. The aim of this study is to evaluate the role of Isotretinoin on immune activation and inflammation.
  Other Names: 13-cis-retinoic acid
  Arms: Isotretinoin Arm

SUMMARY:
This phase II study was done in HIV-infected participants on antiretroviral therapy to evaluate the effects of isotretinoin (a drug that is approved for use in the treatment of severe acne) on the immune system. The immune system helps the body fight infections. When the immune system is not working well, one may be at greater risk for diseases that are common in aging, like heart disease, weaker bones, and kidney disease.

DETAILED DESCRIPTION:
Isotretinoin was administered to participants in the Isotretinoin arm at approximately 0.5 mg/kg PO once daily for 4 weeks, then increased to approximately 1.0 mg/kg PO once daily for 12 weeks. Follow-up continues to week 28 to evaluate the duration of effect. Randomization was stratified by willingness to participate in the gut biopsy substudy, A5330s. The study population included HIV-1 infected adults whose virus was suppressed on ART, excluding women of child bearing potential.

ELIGIBILITY:
Inclusion Criteria:

- HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 antigen, plasma HIV-1 RNA viral load.

NOTE: The term "licensed" refers to a US FDA-approved kit, which is required for all IND studies.

CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (eg, indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.

* Receiving ART therapy for at least 12 months prior to study entry.
* No plans to change the ART regimen in the 6 months after study entry.
* HIV-1 RNA below the lower limit of detection using an FDA-approved assay obtained within 30 days prior to study entry by any laboratory that has a CLIA certification or its equivalent (eg, <50 copies/mL on Roche Amplicor HIV-1 Monitor assay, <75 copies/mL on the Versant HIV-1 RNA assay by branched DNA, <40 copies/mL on the Abbott m2000sp/m2000rt real-time PCR test, < 20 copies/mL on the COBAS AmpliPrep/TAQMAN HIV-1 assay).
* All measurements of HIV-1 RNA within the 12 months prior to study entry must be below the limit of detection with the following exception:

NOTE A: 1 viral blip (<200 copies/mL) is permitted if it is preceded and followed by viral loads below the limits of detection.

NOTE B: The virologic assay must have a lower limit of detection of ≤ 75 copies/mL.

* CD4+ cell count <350 cells/mm3 obtained at screening within 30 days prior to entry at any laboratory that has a CLIA (Clinical Laboratory Improvement Amendments) certification or its equivalent.
* The following laboratory values obtained within 30 days prior to entry by any laboratory that has a CLIA certification or its equivalent:

  1. Hemoglobin A1c (HgbA1c) levels ≤ 6.5%
  2. Hemoglobin ≥ 9.0 g/dL
  3. Platelet count ≥ 50,000/mm3
  4. Creatinine ≤1.5 mg/dl
  5. CrCl ≥ 60 mL/min, calculated by the Cockcroft-Gault method
  6. Aspartate aminotransferase (AST) (SGOT) ≤1.5x upper limit of normal (ULN)
  7. Alanine aminotransferase (ALT) (SGPT) ≤1.5x ULN
  8. Serum lipase ≤1.5x ULN
  9. Fasting triglyceride level ≤200 mg/dL
  10. Fasting glucose <126mg/dL
* Karnofsky performance score >/=70 within 30 days prior to entry.
* Men and post-menopausal females aged ≥ 18 years and ≤ 80 years at entry.

Note: Post-menopausal is defined as having either:

1. Appropriate medical documentation (see note) of prior complete bilateral oophorectomy (i.e., surgical removal of the ovaries, resulting in "surgical menopause" and occurring at the age at which the procedure was performed), OR
2. Permanent cessation (12 consecutive months or more of amenorrhea) of previously occurring menses as a result of ovarian failure with documentation of hormonal deficiency by a certified healthcare provider (i.e., "spontaneous menopause").

Hormonal deficiency should be properly documented (see note) in the case of suspected spontaneous menopause as follows:

1. If age >54 years and with the absence of normal menses: Serum FSH (Follicle Stimulating Hormone) level elevated to within the post-menopausal range based on the laboratory reference range where the hormonal assay is performed.
2. If age ≤ 54 years and with the absence of normal menses: Negative serum or urine HCG with concurrently elevated serum FSH (follicle stimulating hormone) level in the post-menopausal range, depressed estradiol (E2) level in the post-menopausal range, and absent serum progesterone level, based on the laboratory reference ranges where the hormonal assays are performed.

NOTE: "Appropriate documentation", and "properly documented" means written documentation or oral communication from a clinician or clinician's staff documented in source documents of an operative report, discharge summary, or

* No active hepatitis B or C infection. NOTE: For subjects who have documentation of prior infection, but no active hepatitis infection, evidence of clearance must be greater than 1 year.
* Ability and willingness of subject to provide informed consent.
* Willingness to adhere to the iPLEDGE program requirements.
* Indication of willingness to participate in the substudy A5330s. NOTE: In the event that 12 or fewer subjects have enrolled into A5330s by the time enrollment in the main study has reached 50% of the accrual target, A5330s enrollment will be required.

Exclusion Criteria:

* Pre-existing diagnosis of diabetes.
* Currently receiving treatment with fibrate, nicotinic acid, tetracycline, fish oil >1g/d, or methotrexate.
* Known active healing fracture or any severe bone disorders. NOTE: does not include healed fractures or history of old fractures.
* Receipt of any of the following medications within 30 days prior to entry: systemic steroids (including intra-articular steroids; inhaled or nasal steroid therapy is permitted), interleukins, systemic interferons (including intra-articular steroid injection; local injection of interferon alpha for treatment of human papilloma virus is permitted), or systemic chemotherapy.
* Known allergy/sensitivity or any hypersensitivity to vitamin A, retinoids, or any of their derivatives.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Acute or serious illness requiring systemic treatment and/or hospitalization within 60 days prior to entry.
* Weight < 40 kg or > 150 kg.
* History of major depression or suicide attempt requiring hospitalization, or psychotic episode requiring medication or hospitalization.
* History of inflammatory bowel disease such as Crohn's disease, or Ulcerative colitis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2014-07-02 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Kwon, MD, PhD, Study Chair — Massachusetts General Hospital; Nina Lin, MD, Study Chair — Harvard Medical School (HMS and HSDM)
Locations (15):
- United States (14):
  - 31788 Alabama CRS, Birmingham, Alabama
  - 601 University of California, Los Angeles CARE Center CRS, Los Angeles, California
  - 801 University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - 101 Massachusetts General Hospital (MGH) CRS, Boston, Massachusetts
  - 107 Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - 2101 Washington University Therapeutics (WT) CRS, St Louis, Missouri
  - 31786 New Jersey Medical School Clinical Research Center CRS, Newark, New Jersey
  - 31787 University of Rochester Adult HIV Therapeutic Strategies Network CRS, Rochester, New York
  - 3201 Chapel Hill CRS, Chapel Hill, North Carolina
  - 3203 Greensboro CRS, Greensboro, North Carolina
  - 2401 Cincinnati CRS, Cincinnati, Ohio
  - 2951 The Miriam Hospital (TMH) ACTG CRS, Providence, Rhode Island
  - 3652 Vanderbilt Therapeutics (VT) CRS, Nashville, Tennessee
  - 31473 Houston AIDS Research Team (HART) CRS, Houston, Texas
- 5401 Puerto Rico AIDS Clinical Trials Unit CRS, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant was enrolled on July 2, 2014. Accrual to the study closed on May 5, 2016, with 15 U.S and Puerto Rico sites registered and enrolled participants
Pre-assignment Details: Participants were randomized 2:1 to Isotretinoin and no study treatment arms. Randomization was stratified by willingness to participate in the gut biopsy substudy, A5330s.
Period: Overall Study
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Started | 50 | 26
Completed | 47 | 26
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Isotretinoin Arm | No Study Treatment Arm | Total
Number analyzed (Participants) | 50 | 26 | 76
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [38 to 55] | 51 [38 to 53] | 49 [38 to 55]
Age, Customized [Count of Participants; unit: Participants]
  18-39 years | 14 | 7 | 21
  40-59 years | 31 | 16 | 47
  >=60 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 46 | 25 | 71
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 18 | 12 | 30
  Non-Hispanic Black | 21 | 9 | 30
  Hispanic (Regardless of Race) | 11 | 5 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  Puerto Rico | 1 | 0 | 1
  United States | 49 | 26 | 75
HIV-1 RNA [Count of Participants; unit: Participants]
  >= Assay lower limit (40 copies/mL) | 0 | 1 | 1
  < Assay lower limit (40 copies/mL) | 50 | 25 | 75
CD4+ Cell Count [Median (Inter-Quartile Range); unit: cells/mm^3] | 549 [299 to 754] | 556 [342 to 781] | 552 [310 to 768]
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 27.1 [23.1 to 29.3] | 26.9 [22.6 to 27.9] | 27.1 [22.9 to 29.2]
CD8+ T-cell Activation Percent [Median (Inter-Quartile Range); unit: percentage of cells] — CD8+ T-cell activation percent is the primary endpoint. Level of CD8+ T-cell activation was determined by measuring the percentage of cells that expressed both the activation marker CD38+ and Human leukocyte antigen (HLA)-DR+.
  Baseline is defined as the average of pre-entry and entry values Population: The primary endpoint is limited to participants who have data for both baseline and week 14/16, (for the Isotretinoin arm) completed treatment (allowing ≤8 missed doses), did not use prohibited medications, and did not experience virologic failure from baseline to week 16.
  percentage of cells
    number analyzed (Participants) | 39 | 26 | 65
    (all) | 13.67 [10.35 to 19.49] | 13.40 [8.43 to 18.56] | 13.66 [9.83 to 19.29]

OUTCOME MEASURES:

1. Primary Outcome: Change in CD8+ T-cell Activation From Baseline to Week 14/16
Description: Level of CD8+ T-cell activation was determined by measuring the percentage of CD8+ T-cells that expressed both the activation marker CD38+ and Human leukocyte antigen (HLA)-DR+. The endpoint is measuring the change from baseline to week 14/16, where baseline is defined as the average of pre-entry and entry, and week 14/16 is defined as the average of week 14 and week 16.
  Change = (week 14/16 - baseline).
Time Frame: baseline, week 14/16
Population: The primary analysis is complete case as-treated, and is limited to participants who:
  * have data for both baseline and week 14/16
  * (for the Isotretinoin arm) completed treatment (allowing ≤8 missed doses)
  * did not use prohibited medications
  * did not experience virologic failure from baseline to week 16
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
percentage of cells | 3.24 [0.77 to 7.75] | 0.52 [-0.41 to 2.86]
Statistical Analysis 1: Comparison: Isotretinoin Arm vs No Study Treatment Arm; Null hypothesis: There is no difference between the two arms in the change in T-cell activation from baseline to week 14/16; Test type: Superiority; p = 0.030, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons

2. Secondary Outcome: Change in CD8+ T-cell Activation
Description: Level of CD8+ T-cell activation was determined by measuring the percentage of CD8+ T-cells that expressed both the activation marker CD38+ and Human leukocyte antigen (HLA)-DR+.
  The endpoint is measuring the change from week 14/16 to week 28 (week 28 - week 14/16) and from baseline to week 28 (week 28 - baseline).
  Baseline is defined as the average of pre-entry and entry, and week 14/16 is defined as the average of week 14 and week 16.
Time Frame: baseline, week 14/16, week 28
Population: The analysis is complete case as-treated, and is limited to participants who:
  * have data for both baseline and week 14/16
  * (for the Isotretinoin arm) completed treatment (allowing ≤8 missed doses)
  * did not use prohibited medications
  * did not experience virologic failure from baseline to week 16
Measure: Median (Inter-Quartile Range); unit: percentage of cells
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
percentage of cells
  Change from week 14/16 to week 28 | -3.58 [-8.45 to 0.35] | -0.91 [-3.40 to 1.49]
  Change from baseline to week 28 | -0.69 [-2.61 to 4.00] | 0.03 [-2.34 to 3.32]

3. Secondary Outcome: Change in sCD14
Description: sCD14 (soluble cluster of differentiation 14) is a marker of gut microbial translocation and monocyte activation.
  The outcome measures are changes in log10 transformed sCD14 from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 pg/mL
  Change from baseline to week 14/16 | 0.02 [-0.03 to 0.10] | -0.02 [-0.06 to 0.05]
  Change from week 14/16 to week 28 | -0.06 [-0.13 to 0.02] | 0.02 [-0.04 to 0.06]
  Change from baseline to week 28 | -0.02 [-0.07 to 0.05] | 0.00 [-0.06 to 0.05]

4. Secondary Outcome: Change in I-FABP
Description: I-FABP (intestinal-fatty acid binding protein) is a marker of intestinal cell damage and turnover.
  The outcome measures are changes in log10 transformed I-FABP from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 pg/mL
  Change from baseline to week 14/16 | -0.03 [-0.14 to 0.10] | 0.04 [-0.05 to 0.17]
  Change from week 14/16 to week 28 | 0.09 [-0.01 to 0.16] | -0.05 [-0.15 to 0.05]
  Change from baseline to week 28 | 0.07 [-0.05 to 0.20] | -0.07 [-0.19 to 0.11]

5. Secondary Outcome: Change in IL-6
Description: IL-6 (Interleukin-6) is a marker of systemic inflammation. The outcome measures are changes in log10 transformed IL-6 from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 pg/mL
  Change from baseline to week 14/16 | 0.10 [-0.02 to 0.19] | -0.04 [-0.11 to 0.05]
  Change from week 14/16 to week 28 | -0.08 [-0.27 to 0.03] | 0.01 [-0.07 to 0.13]
  Change from baseline to week 28 | 0.02 [-0.14 to 0.17] | -0.01 [-0.14 to 0.16]

6. Secondary Outcome: Change in hsCRP
Description: hsCRP (high-sensitivity C-reactive protein) is a marker of inflammation. Change in log10 transformed hsCRP from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 ng/mL
  Change from baseline to week 14/16 | 0.20 [-0.07 to 0.32] | -0.08 [-0.21 to 0.19]
  Change from week 14/16 to week 28 | -0.24 [-0.52 to -0.06] | 0.11 [-0.06 to 0.31]
  Change from baseline to week 28 | -0.09 [-0.39 to 0.18] | -0.05 [-0.15 to 0.29]

7. Secondary Outcome: Change in sTNF-r1
Description: sTNF-r1 (soluble tumour necrosis alpha receptor 1) is a marker of inflammation. Change in log10 transformed sTNF-r1 from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 pg/mL
  Change from baseline to week 14/16 | 0.00 [-0.02 to 0.03] | 0.01 [-0.03 to 0.05]
  Change from week 14/16 to week 28 | 0.00 [-0.04 to 0.02] | 0.00 [-0.03 to 0.04]
  Change from baseline to week 28 | 0.00 [-0.04 to 0.03] | 0.02 [-0.03 to 0.04]

8. Secondary Outcome: Change in sTNF-r2
Description: sTNF-r2 (soluble tumour necrosis alpha receptor 2) is a marker of inflammation. Change in log10 transformed sTNF-r2 from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 pg/mL
  Change from baseline to week 14/16 | 0.03 [-0.02 to 0.07] | 0.01 [-0.02 to 0.05]
  Change from week 14/16 to week 28 | -0.02 [-0.08 to 0.03] | 0.00 [-0.04 to 0.04]
  Change from baseline to week 28 | 0.00 [-0.03 to 0.04] | 0.02 [-0.02 to 0.06]

9. Secondary Outcome: Change in D-dimer
Description: D-dimer (or D dimer) is a marker of coagulation activation. Change in log10 transformed D-dimer from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 ng/mL
  Change from baseline to week 14/16 | 0.10 [0.01 to 0.20] | 0.02 [-0.05 to 0.15]
  Change from week 14/16 to week 28 | -0.04 [-0.22 to 0.03] | 0.00 [-0.04 to 0.07]
  Change from baseline to week 28 | 0.01 [-0.07 to 0.14] | 0.09 [-0.05 to 0.14]

10. Secondary Outcome: Change in TF
Description: TF (Tissue Factor) is a marker of Coagulation. Change in log10 transformed TF from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 pg/mL
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 pg/mL
  Change from baseline to week 14/16 | -0.01 [-0.02 to 0.03] | 0.01 [-0.02 to 0.05]
  Change from week 14/16 to week 28 | 0.00 [-0.07 to 0.03] | 0.01 [0.00 to 0.04]
  Change from baseline to week 28 | -0.02 [-0.06 to 0.03] | 0.03 [0.01 to 0.07]

11. Secondary Outcome: Change in sCD163
Description: sCD163 (soluble CD 163) is a marker of macrophage activation Change in log10 transformed sCD163 from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: log10 ng/mL
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 ng/mL
  Change from baseline to week 14/16 | 0.15 [0.04 to 0.22] | -0.01 [-0.04 to 0.12]
  Change from week 14/16 to week 28 | -0.14 [-0.19 to -0.05] | -0.01 [-0.08 to 0.05]
  Change from baseline to week 28 | -0.02 [-0.10 to 0.15] | 0.04 [-0.08 to 0.21]

12. Secondary Outcome: Change in CD4+ T-cell Count
Description: Change in peripheral total CD4 cell count from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: cells/mm^3
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
cells/mm^3
  Change from baseline to week 14/16: number analyzed (Participants) | 38 | 26
  Change from baseline to week 14/16 | 17 [-35 to 43] | -39 [-124 to 19]
  Change from week 14/16 to week 28: number analyzed (Participants) | 38 | 25
  Change from week 14/16 to week 28 | 31 [-10 to 75] | 21 [-31 to 81]
  Change from baseline to week 28: number analyzed (Participants) | 39 | 25
  Change from baseline to week 28 | 27 [-18 to 89] | -14 [-76 to 30]

13. Secondary Outcome: Change in Cell-associated HIV-1 RNA
Description: Cell-associated HIV-1 RNA in blood from baseline to week 14/16(week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
  For cell-associated HIV-1 RNA results below the assay limit, the lowest value of the sample was imputed to these results (1.32 log10 copies/10^6 CD4 cells).
  Since there are only a few results below the assay limit, it is still reasonable to summarize the absolute changes for cell-associated HIV-1 RNA, where changes were calculated based on the imputed values (described above) for below assay limit results.
Time Frame: baseline, week 14/16, week 28
Population: The analysis is complete case as-treated, and is limited to participants who:
  * have data for both baseline and week 14/16
  * (for the Isotretinoin arm) completed treatment (allowing ≤8 missed doses)
  * did not use prohibited medications
  * did not experience virologic failure from baseline to week 16
  * have cell-associated HIV-1 RNA data
Measure: Median (Inter-Quartile Range); unit: log10 copies/million CD4 cells
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 37 | 26
log10 copies/million CD4 cells
  Change from baseline to week 14/16: number analyzed (Participants) | 35 | 26
  Change from baseline to week 14/16 | -0.09 [-0.32 to 0.24] | -0.02 [-0.22 to 0.25]
  Change from week 14/16 to week 28: number analyzed (Participants) | 33 | 24
  Change from week 14/16 to week 28 | -0.03 [-0.28 to 0.22] | -0.20 [-0.51 to 0.04]
  Change from baseline to week 28: number analyzed (Participants) | 37 | 24
  Change from baseline to week 28 | -0.08 [-0.28 to 0.13] | -0.18 [-0.46 to 0.12]

14. Secondary Outcome: Cell-associated HIV-1 DNA
Description: Cell-associated HIV-1 DNA in blood at baseline, week 14/16, and week 28. Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
  For cell-associated HIV-1 DNA results below the assay limit, the lowest value of the sample was imputed to these results and considered lowest ranks (1.62 log10 copies/10^6 CD4 cells).
  It was originally planned to summarize the absolute changes for cell-associated HIV-1 DNA. However, since there are many results below limit of detection, analyzing the absolute changes would be inappropriate in this case.
  Instead, the baseline, week 14/16, and week 28 levels were summarized.
Time Frame: baseline, week 14/16, week 28
Population: The analysis is complete case as-treated, and is limited to participants who:
  * have data for both baseline and week 14/16
  * (for the Isotretinoin arm) completed treatment (allowing ≤8 missed doses)
  * did not use prohibited medications
  * did not experience virologic failure from baseline to week 16
  * have cell-associated HIV-1 DNA data
Measure: Median (Inter-Quartile Range); unit: log10 copies/million CD4 cells
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
log10 copies/million CD4 cells
  baseline | 2.55 [2.03 to 2.99] | 2.72 [2.39 to 2.94]
  week 14/16: number analyzed (Participants) | 37 | 26
  week 14/16 | 2.52 [2.25 to 2.79] | 2.66 [2.23 to 2.88]
  week 28: number analyzed (Participants) | 38 | 25
  week 28 | 2.64 [1.78 to 2.95] | 2.55 [2.21 to 2.82]

15. Secondary Outcome: Change in Treg Frequency (%FoxP3+/CD25hi+/CD39+/CD127-(CD4+))
Description: Treg (T Regulatory) Cells are a subpopulation of T cells which modulate the immune system.
  The outcome measure is the change in percent FoxP3+/CD25hi+/CD39+/CD127-(CD4+) from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of CD4 cells
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
percentage of CD4 cells
  Change from baseline to week 14/16 | 0.00 [-0.46 to 0.20] | -0.03 [-0.29 to 0.25]
  Change from week 14/16 to week 28: number analyzed (Participants) | 38 | 26
  Change from week 14/16 to week 28 | 0.00 [-0.28 to 0.26] | 0.02 [-0.11 to 0.21]
  Change from baseline to week 28: number analyzed (Participants) | 38 | 26
  Change from baseline to week 28 | -0.03 [-0.36 to 0.09] | 0.11 [-0.26 to 0.26]

16. Secondary Outcome: Change in Th17 Frequency (%IFNg-/IL17+(CD161+/CCR6+))
Description: Th17 (T-helper 17) cells are a subset of pro-inflammatory T helper cells defined by their production of interleukin 17 (IL-17).
  The outcome is the change in percent IFNg-/IL17+(CD161+/CCR6+) from baseline to week 14/16 (week 14/16 - baseline), from week 14/16 to week 28 (week 28 - week 14/16), and from baseline to week 28 (week 28 - baseline).
  Levels measured at pre-entry and entry were averaged for baseline, levels measured at week 14 and week 16 were averaged for week 14/16.
Time Frame: baseline, week 14/16, week 28
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: percentage of CD161+/CCR6+ cells
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 39 | 26
percentage of CD161+/CCR6+ cells
  Change from baseline to week 14/16 | -0.04 [-0.42 to 0.14] | 0.01 [-0.31 to 0.54]
  Change from week 14/16 to week 28: number analyzed (Participants) | 38 | 26
  Change from week 14/16 to week 28 | 0.02 [-0.33 to 0.28] | -0.07 [-0.41 to 0.18]
  Change from baseline to week 28: number analyzed (Participants) | 38 | 26
  Change from baseline to week 28 | -0.05 [-0.50 to 0.14] | -0.01 [-0.85 to 0.52]

17. Secondary Outcome: Pharmacokinetics - Endogenous Levels of Retinoid Metabolites for Isotretinoin Arm
Description: Isotretinoin Arm (Arm A) only. Endogenous retinoid metabolites are defined as the average concentrations of Retinol, and Total Retinyl Ester from weeks 0, 20, and 28.
Time Frame: weeks 0, 20, 28
Population: Included only Isotretinoin arm participants who were on Isotretinoin for 8 weeks of more.
Measure: Median (Inter-Quartile Range); unit: nmol/mL
Arm/Group | Isotretinoin Arm
Number analyzed (Participants) | 39
nmol/mL
  Retinol | 2.4 [1.8 to 2.7]
  Total Retinyl Ester | 0.5 [0.4 to 0.6]

18. Secondary Outcome: Pharmacokinetics - Steady-state Trough Concentrations of Isotretinoin for Isotretinoin Arm
Description: Isotretinoin arm (Arm A) only, steady-state trough concentrations of Isotretinoin is defined as the average of 'eligible' concentrations at weeks 8, 12, and 16, where 'eligible' means the time from the previous dose to the blood draw of the sample must have been in the 14-to-30 hour range, and the participant must have taken at least 3 doses in the prior 4 days.
Time Frame: weeks 8, 12, 16
Population: Included only Isotretinoin arm participants who were on Isotretinoin for 8 weeks of more and have steady state troughs available.
Measure: Median (Inter-Quartile Range); unit: pmol/mL
Arm/Group | Isotretinoin Arm
Number analyzed (Participants) | 30
pmol/mL
  All | 205 [152 to 263]
  With EFV: number analyzed (Participants) | 7
  With EFV | 228 [120 to 265]
  No EFV: number analyzed (Participants) | 23
  No EFV | 202 [152 to 241]

19. Secondary Outcome: Pharmacokinetics - Trough Concentrations of TDF for Isotretinoin Arm
Description: Isotretinoin arm (Arm A) only, trough concentrations of TDF (Tenofovir) is defined as the average of 'eligible' concentrations, where 'eligible' means the time from the previous dose to the blood draw of the sample must have been in the 20-to-28 hour range, and the participant must have taken at least 3 doses in the prior 4 days.
  TDF trough during Isotretinoin administration is the average of 'eligible' concentrations from weeks 8, 12, and 16; TDF trough without Isotretinoin administration is the average of 'eligible' concentrations from weeks 0 and 20.
  (Week 28 data is not available.)
Time Frame: weeks 0, 8, 12, 16, 20
Population: Included only Isotretinoin arm participants who were on TDF and on Isotretinoin for 8 weeks of more, and with available TDF trough.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Isotretinoin Arm
Number analyzed (Participants) | 15
ng/mL
  With Isotretinoin | 82 [52 to 107]
  Without Isotretinoin | 63 [46 to 87]

20. Secondary Outcome: Pharmacokinetics - 12-hour Levels of EFV for Isotretinoin Arm
Description: Isotretinoin arm (Arm A) only, 12-hour levels of EFV (Efavirenz) is defined as the average of 'eligible' concentrations, where 'eligible' means the time from the previous dose to the blood draw of the sample must have been in the 9-to-15 hour range, and the participant must have taken at least 3 doses in the prior 4 days.
  EFV trough during Isotretinoin administration is the average of 'eligible' concentrations from weeks 8, 12, and 16; EFV trough without Isotretinoin administration is the average of 'eligible' concentrations from weeks 0 and 20.
  (Week 28 data is not available.)
Time Frame: weeks 0, 8, 12, 16, 20
Population: Included only Isotretinoin arm participants who were on EFV and on Isotretinoin for 8 weeks of more, and with available EFV 12-hour levels.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Isotretinoin Arm
Number analyzed (Participants) | 11
ng/mL
  With Isotretinoin | 2607 [1648 to 4343]
  Without Isotretinoin | 2665 [1849 to 3421]

21. Secondary Outcome: Primary Targeted Adverse Events
Description: Targeted events for A5325 include: events that meet the International Conference on Harmonization (ICH) definitions for a serious adverse event, post-entry signs/symptoms and laboratory abnormalities of Grade ≥3 or that lead to a change in treatment regardless of grade, and any diagnoses.
Time Frame: from study entry to end of study (week 28)
Population: all enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Isotretinoin Arm | No Study Treatment Arm
Number analyzed (Participants) | 50 | 26
Participants | 18 | 6

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) reported from study enrollment until study completion at 28 weeks
Description: Expedited adverse event (EAE) reporting followed the Division of AIDS (DAIDS) EAE Manual under the SAE Reporting Category and including fetal losses. Events were graded (1=mild, 2=moderate, 3=severe, 4=life-threatening, 5=death) according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Version 1.0, Clarification Aug 2009.
Groups:
- Isotretinoin: Participants received Isotretinoin at approximately 0.5 mg/kg orally once daily for 4 weeks, then increased to approximately 1.0 mg/kg orally once daily for 12 weeks.
- No Study Treatment: No Isotretinoin treatment
Arm/Group | Isotretinoin | No Study Treatment
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/26
Serious Adverse Events (participants affected / at risk) | 2/50 | 0/26
Other Adverse Events (participants affected / at risk) | 41/50 | 18/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Isotretinoin (N=50) | No Study Treatment (N=26)
Meningitis viral (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Isotretinoin (N=50) | No Study Treatment (N=26)
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 4
Aspartate aminotransferase increased (Investigations) | 0 | 3
Blood alkaline phosphatase increased (Investigations) | 3 | 2
Blood bicarbonate decreased (Investigations) | 3 | 1
Blood bilirubin increased (Investigations) | 7 | 2
Blood cholesterol increased (Investigations) | 20 | 11
Blood creatinine increased (Investigations) | 3 | 2
Blood glucose decreased (Investigations) | 3 | 1
Blood glucose increased (Investigations) | 10 | 5
Blood potassium decreased (Investigations) | 3 | 2
Blood sodium decreased (Investigations) | 3 | 1
Lipase abnormal (Investigations) | 3 | 2
Low density lipoprotein increased (Investigations) | 18 | 8
Neutrophil count decreased (Investigations) | 2 | 2
Platelet count decreased (Investigations) | 2 | 2
Headache (Nervous system disorders) | 3 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.